CLINICAL TRIAL: NCT05018286
Title: An Open-label Extension Trial to Evaluate the Long-term Safety of Apraglutide in Short Bowel Syndrome.
Brief Title: Open-label Extension Trial to Evaluate the Long-term Safety of Apraglutide in Short Bowel Syndrome.
Acronym: STARS extend
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: VectivBio AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TA799-012
Record Dates: First submitted 2021-07-06; First posted 2021-08-24 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Short Bowel Syndrome
Keywords: Short Bowel Syndrome; SBS; Intestinal Failure; SBS-IF
MeSH Terms: conditions — Short Bowel Syndrome; Intestinal Failure | interventions — apraglutide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Apraglutide subcutaneous (SC) injections, once weekly (Experimental): Peptide analogue of Glucagon-like Peptide 2 (GLP-2)
  Interventions: Drug: Apraglutide

INTERVENTIONS:
Drug: Apraglutide — Apraglutide is a synthetic peptide analogue of GLP-2 under development for treatment of SBS-IF, which acts as a full agonist at the GLP-2 receptor with in vitro potency and selectivity comparable with native GLP-2

SUMMARY:
The primary objective of the trial is to assess long-term safety and tolerability of apraglutide in subjects with SBS-IF.

DETAILED DESCRIPTION:
This is an international, multicenter, open label extension trial to collect further safety, tolerability, efficacy, durability, and clinical outcomes of apraglutide once weekly adminstration, for up to 208 weeks or until apraglutide is commercially available in the country, whichever comes first. Eligible subjects would be those who were trial subjects of TA799-007 or TA799-013 trials.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females with a diagnosis of SBS-IF secondary to surgical resection of the small intestine, with Colon-in-Continuity (CIC) or stoma, who were trial subjects of parent trials TA799-007 or TA799-013
2. Able to give informed consent and agree to follow the details of participation as outlined in the protocol.

Exclusion Criteria:

1. Subject not capable of understanding or not willing to adhere to the trial visit schedules and other protocol requirements.
2. Any other reason judged not eligible by the Investigator.
3. Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AE) | From baseline to week 208
  System organ class, frequency and severity
Clinical chemistry | From baseline to week 208
  Clinical Chemistry panel of analytes will be examined for clinically significant changes.
Hematology | From baseline to week 208
  Hematology panel of analytes will be examined for clinically significant changes.
Hemostasis | From baseline to week 104
  Hemostasis INR will be examined for clinically significant changes.
Urinalysis | From baseline to week 208
  Urinanalysis panel of analytes will be examined for clinically significant changes.
Occurrence of clinically relevant changes in vital signs | From baseline to week 208
  * Systolic and diastolic blood pressure in mmHg will be examined for clinically significant changes.
  * Heart rate in Beats per Minute (BPM) will be examined for clinically significant changes.
Occurrence of clinically relevant changes in electrocardiogram | From baseline to week 208
  ECG; intervals and rhythm

SECONDARY OUTCOMES:
Change from baseline in PS volume | From baseline to week 208
Change from baseline in PS frequency | From baseline to week 208
  Change in PS days/week from baseline to week 104
Clinically significant changes in PS total energy | From baseline to week 208
  Units: kcal
Change from baseline in PS infusion time | From baseline to week 208
Percentage of subjects reaching enteral autonomy | From baseline to week 104
Change from baseline in body weight | From baseline to week 104
  Units: kg
Change from baseline on the Patient Global Impression of Severity (PGIS) | From baseline to week 104
Change from baseline on the Pittsburgh Sleep Quality Inventory (PSQI) | From baseline to week 208
Change from baseline on the Patient Global Impression of Change (PGIC) | From baseline to week 208
Changes from baseline on Patient Global Impression of Treatment Satisfaction (PGI-TS) | From baseline to week 208
Changes from baseline on Patient Global Impression of Satisfaction with Parenteral Support (PGI-SPS) | From baseline to week 208
Changes from baseline on Patient Global Impression of Parenteral Support Impact (PGI-PSI) | From baseline to week 208
Change from baseline on the Short Form (36) Health Survey (SF-36) | From baseline to week 208
Change from baseline on the EuroQoL-5 dimension -5 level survey (EQ-5D-5L) | From baseline to week 208

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Masior, Study Director — VectivBio AG
Locations (66):
- United States (13):
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Gastroenterology Group of Naples, Naples, Florida
  - Northwestern University - Chicago, Chicago, Illinois
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Mount Sinai Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Washington Medical Center, Seattle, Washington
- University Hospital Fundacion Favaloro, Buenos Aires, Argentina
- Belgium (2):
  - University Hospital Brussels, Brussels
  - UZ Leuven, Leuven
- Czechia (6):
  - University Hospital Brno, Brno
  - University Hospital Hradec Kralove, Hradec Králové
  - Hospital Novy Jicin, Nový Jičín
  - University Hospital Plzen, Pilsen
  - University Hospital Kralovske Vinohrady, Prague
  - General University Hospital in Prague, Prague
- Rigshospitalet - University Hospital Copenhagen, Department of Intestinal Failure and Liver Diseases, Copenhagen, Denmark
- France (6):
  - Beaujon Hospital, Clichy
  - South Lyon Hospital Center, Lyon
  - Nantes University Hospital Center - Hotel Dieu Hospital, Nantes
  - Nice University Hospital Center - Archet 1 Hospital, Nice
  - Hôpital Haut-Lévèque, Pessac
  - Brabois Adults Hospital, Vandœuvre-lès-Nancy
- Germany (5):
  - Charite - University Hospital Berlin, Berlin
  - University Hospital Bonn, Bonn
  - Asklepios Clinic St. Georg, Hamburg
  - University Hospital Heidelberg, Heidelberg
  - University Hospital Muenster, Münster
- Hungary (4):
  - Szent Imre University Teaching Hospital, Department of Gastroenterology, Budapest
  - Central Hospital of Northern Pest - Military Hospital, Budapest
  - Semmelweis University, Budapest
  - University of Szeged, Szeged
- Israel (2):
  - Rambam Health Care Campus, Institute of Gastroenterology, Haifa
  - Chaim Sheba Medical Center, Tel Litwinsky
- Italy (3):
  - Polyclinic S. Orsola-Malpighi, Bologna
  - University Polyclinic Foundation "Agostino Gemelli" - IRCCS, Rome
  - City of Health and Science of Turin, Turin
- Japan (5):
  - Yokohama City University Medical Center, Kanagawa
  - Yokohama Municipal Citizen's Hospital, Kanagawa
  - Osaka University Hospital, Osaka
  - Tohoku University Hospital, Sendai
  - JCHO Tokyo Yamate Medical Center, Tokyo
- More og Romsdal Hospital Trust - Alesund Hospital, Ålesund, Norway
- Poland (5):
  - Stadmedica, Non-Public Healthcare Facility, Bydgoszcz
  - COPERNICUS Limited Liability Company, Nutrition Outpatient Clinic for Adults, Gdansk
  - M. Pirogow Provincial Specialized Hospital, Lodz
  - Gastromed Poland Sp. z o.o., Lublin
  - Stanley Dudrick Multispecialty Hospital, Skawina
- South Korea (3):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (3):
  - University General Hospital Gregorio Maranon, Madrid
  - University Hospital 12 de Octubre, Madrid
  - University Hospital Virgen del Rocio (HUVR), Seville
- Sahlgrenska University Hospital, Sahlgrenska Intestinal Failure and Transplant Centre, Gothenburg, Sweden
- Far Eastern Memorial Hospital, New Taipei City, Taiwan
- United Kingdom (4):
  - St Mark's Hospital, Harrow
  - Royal London Hospital, London
  - University College Hospital, London
  - Northern Care Alliance NHS Foundation Trust, Salford